CLINICAL TRIAL: NCT06485401
Title: An Phase I, Open-label, Multi-center, Parallel, Single Oral Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of ADC189 in Subjects With Hepatic Impairment (Child-Pugh A and B) Compared With Subjects With Normal Hepatic Function
Brief Title: To Compare the Safety and PK/ PD Characteristics of ADC189 Between Hepatic Impairment and Normal Hepatic Function Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiaxing AnDiCon Biotech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-ADC189-I-001
Record Dates: First submitted 2024-06-15; First posted 2024-07-03 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-06

CONDITIONS: Influenza Type A; Influenza Type B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ADC189 to Child-Pugh Class A (Experimental): Subjects with Child-Pugh Class A received a single dose once of ADC189 (45 mg/1 tablet).
  Interventions: Drug: ADC189
- ADC189 to normal haptic function (A) (Experimental): Healthy subjects who marched with Group "Child-Pugh Class A", that received a single dose of ADC189 (45 mg/1 tablet).
  Interventions: Drug: ADC189
- ADC189 to Child-Pugh Class B (Experimental): Subjects with Child-Pugh Class B received a single dose once of ADC189 (45 mg/1 tablet).
  Interventions: Drug: ADC189
- ADC189 to normal haptic function (B) (Experimental): Healthy subjects who marched with Group "Child-Pugh Class B", that received a single dose of ADC189 (45 mg/1 tablet).
  Interventions: Drug: ADC189

INTERVENTIONS:
Drug: ADC189 — 45 mg per tablet, oral administration, single dose.

SUMMARY:
This study aims to evaluate the pharmacokinetics, pharmacodynamics, safety, and tolerability of ADC189 in subjects with hepatic impairment compared with subjects with normal hepatic function.

DETAILED DESCRIPTION:
The evaluation of ADC189/ADC189-I07 in mild hepatic insufficiency (Child-Pugh A), moderate hepatic insufficiency (Child-Pugh B) the pharmacokinetic characteristics in subjects, compared with normal liver function subjects, which matched by sex, age, and BMI, in order to provide a scientific basis for a reasonable dosage in patients with liver dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 1) The subjects fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign a written informed consent, and can complete the entire trial process according to the requirements of the trial.
* 2) Age 18-75 years old (including the boundary value), both male and female.
* 3) The body weight of male subjects was ≥50 kg, the body weight of female subjects was ≥45 kg, and the body mass index (BMI) was within the range of 18.0~30.0 kg/m².

Exclusion Criteria:

* 1) Known allergic history to test drug components, or allergic constitution, or history of allergic diseases.
* 2) Have malignant tumors, or have a history of malignant tumors within 5 years prior to screening.
* 3) Patients with severe infection, trauma, gastrointestinal surgery or other major surgical operations within 4 weeks before screening.
* 4) eGFR (CKD-EPI Cr) <60mL/min/1.73m2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Cmax of ADC189/ADC189-I07 | 15 days
AUClast of ADC189/ADC189-I07 | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No